CLINICAL TRIAL: NCT01655238
Title: Have NCH Obesity Guidelines Made an Impact? Differences in Anesthetizing the Obese Child in Outpatient Sites Versus Main OR at NCH.
Brief Title: Obesity Guidelines for Outpatient Surgery
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Vidya Raman, Director of Preoperative Assessment Testing, Nationwide Children's Hospital
Other Study IDs: IRB12-00324
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 95-99% BMI ASC: Patients having a BMI between 95-99% who are seen in the ambulatory surgery centers.
  Interventions: Other: BMI
- 95-99% BMI NCH main OR: Patients having a BMI between 95-99% who are seen in the main operating rooms.
  Interventions: Other: BMI
- >99% BMI NCH main OR: Patients having a BMI >99% who are seen in the main operating rooms.
  Interventions: Other: BMI

INTERVENTIONS:
Other: BMI — Screening guideline to assess body mass index.

SUMMARY:
The investigators are concerned about anesthetizing obese children in outpatient locations in case they need prolonged stay, increased respiratory interventions, or need for post-operative narcotics. The investigators will be using a screening guideline to help us determine the higher risk child based on BMI and co-morbid conditions. The investigators will also be doing a retrospective chart review of 300 patients with BMI 95% and looking at various factors during the operative and post-operative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients 95% or over BMI having outpatient surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Obese patients
Sampling Method: Non-Probability Sample
Enrollment: 1327 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Length of stay | 1 week

SECONDARY OUTCOMES:
Number of subjects with respiratory complications | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Vidya Raman, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Smith HL, Meldrum DJ, Brennan LJ. Childhood obesity: a challenge for the anaesthetist? Paediatr Anaesth. 2002 Nov;12(9):750-61. doi: 10.1046/j.1460-9592.2002.00781.x. PMID 12519133
- [Background] Nafiu OO, Reynolds PI, Bamgbade OA, Tremper KK, Welch K, Kasa-Vubu JZ. Childhood body mass index and perioperative complications. Paediatr Anaesth. 2007 May;17(5):426-30. doi: 10.1111/j.1460-9592.2006.02140.x. PMID 17474948